CLINICAL TRIAL: NCT07089225
Title: A Pilot Companion Cancer Cohort Study to the Wake Forest COSMIC Study (WF-2304) in Patients Reporting Cannabis Use Followed With an Application-Based Cannabis Journal
Brief Title: A Study in Patients Reporting Cannabis Use Followed With an Application-Based Cannabis Journal
Acronym: COSMIC- Releaf
Status: Not yet recruiting | Type: Observational
Sponsor: Scot Remick (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Scot Remick, Oncology Research and Education Principal, MaineHealth
Organization: MaineHealth (Other)
Other Study IDs: 20250219.1100; 5UG1CA189824 (NIH)
Record Dates: First submitted 2025-07-15; First posted 2025-07-28 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is being done because there is a significant lack of data on the use of cannabis amongst cancer patients. The investigators believe that the collection of this data will help researchers and clinicians better understand the needs and the impact of cannabis use in this specific patient population.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years of age or older and able to give verbal informed consent to participate.
* Patients must be able to speak, read and understand English.
* Patients must report use of cannabis at time of study participation.
* Patients must have access to internet and ability to download Releaf™ App (MoreBetter, Ltd.) to a smartphone or tablet and must use Releaf™ App (MoreBetter, Ltd.) for cannabis journaling.
* Patients must be able to send and receive text messages, and be able to interact with web-pages on smartphone or tablet.
* There are 2 scenarios that patients are eligible for participation, and are listed below:

  1. Patients must have a cancer diagnosis for which they are receiving active therapy defined as follows:

     * Surgery - must be within a 30-day pre- and/or post-operative (peri-operative) window if single modality of care. Patients must be 18 years of age or older and able to give verbal informed consent to participate.
     * Radiation - must be within a 30-day pre- (simulation planning phase) and/or post-radiation window if single modality of care.
     * Any anticancer systemic therapy including hormonal, biologic, targeted, and/or cytotoxic chemotherapy. Understandably, numerous patients recruited under surgery and/or radiation will receive systemic therapy as part of combined modality therapy, which is permissible. Regardless, all details regarding cancer diagnosis, stage, and treatment will be collected from the EMR, which will be detailed in the informed consent document.
  2. Any patient in follow-up by their primary oncology care provider and/or AYA and cardio-oncology survivorship clinic(s).
* All patients must be treated within the MHCCN thus ensuring access to clinical data in our system-wide EMR (Epic).
* Patients must obtain their cannabis either from a medical-use store, adult-use (recreational) store or both. Patients must obtain cannabis ONLY from medical/recreational stores. Illicit (or homegrown) sources are strictly prohibited.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Oncology patients, receiving active therapy or in follow up following active therapy, and treated within the MaineHealth Cancer Care Network (MHCCN).
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cannabis Use | Enrollment + 6 months
  In patients who report using cannabis, investigators will measure frequency and dose of cannabis and cannabinoid use, purpose of use (i.e., seeking recreational vs. medicinal effects), type (e.g., flower, concentrate, edibles), route of administration (e.g., smoking, vaping, ingestion, tincture, oil), psychoactive and non-psychoactive content (THC vs. CBD/CBG/CBN content in product), and products sources (from medical dispensaries and/or regulated adult-use stores).

SECONDARY OUTCOMES:
Patient Reported Symptoms | Enrollment + 6 months
  Investigators will measure patient-reported helpful and adverse effects of cannabis and cannabinoid use among cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Scot Remick, MD, Principal Investigator — MaineHealth